CLINICAL TRIAL: NCT06931600
Title: Blinding Integrity Following Multiple Sessions of Simulated or Genuine High Velocity, Low Amplitude (HVLA) Manual Chiropractic Adjustments: a Pilot Study
Brief Title: Simulated vs Genuine Manual Chiropractic Adjustments
Acronym: SHA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: I-0032
Record Dates: First submitted 2025-03-28; First posted 2025-04-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Subluxation
Keywords: randomized; sham-controlled; chiropractic; blinding; gait analysis; impedance cardiography; movement parameters; electrocardiography; autonomic nervous system; Heart Rate Variability
MeSH Terms: conditions — Joint Dislocations | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: randomized, sham-controlled, pilot study
Who Masked: Participant, Outcomes Assessor
Masking Description: Lab coordinator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulated/sham (Sham Comparator): 30 individuals receiving simulated/sham chiropractic interventions
  Interventions: Procedure: Sham adjustment
- Genuine/real (Experimental): 30 individuals receiving genuine/real chiropractic interventions
  Interventions: Procedure: Chiropractic adjustment

INTERVENTIONS:
Procedure: Sham adjustment — Two manual high velocity, low amplitude (HVLA) simulated/sham chiropractic interventions in the cervical, thoracic, and/or lumbopelvic regions
  Arms: Simulated/sham
Procedure: Chiropractic adjustment — Two manual high velocity, low amplitude (HVLA) genuine/real chiropractic interventions in the cervical, thoracic, and/or lumbopelvic regions
  Arms: Genuine/real

SUMMARY:
Our primary aim with this trial is to measure participant blinding following two simulated/sham or genuine/real high velocity, low amplitude (HVLA) manual chiropractic adjustments to assess if participants are able to identify their un-disclosed treatment group. Our secondary aims with this trial are to utilize electrocardiography (ECG), impedance cardiography (ICG), and gait analysis before either treatment session and after both treatment sessions to assess if there are any changes with the participants' measurements before and after a sham or genuine HVLA chiropractic treatment.

DETAILED DESCRIPTION:
The primary aim of this trial is to assess blinding following simulated/sham or genuine/real high velocity, low amplitude (HVLA) manual chiropractic adjustments. Briefly, 60 eligible participants will be randomized (1:1 ratio) to receive two sessions of either simulated/sham or genuine/real chiropractic spinal adjustments with a 1 week washout between each treatment. The participants will be given a brief survey immediately following their first and second sessions, as well as immediately prior to the second session. This survey captures their perceptions and experiences regarding the intervention they received. The participants will also complete a pre- and post-electrocardiogram (ECG), impedance cardiography (ICG), and gait analysis. The participant will wear electrical diodes to assess ECG and ICG. Additional sensors will be placed on the participant to assess gait patterns while walking on a treadmill.

ELIGIBILITY:
* No history of stroke or transient ischemic attack or current symptoms including: Dizziness or vertigo; Tinnitus (ringing in the ears); Visual, sensory, or motor disturbances
* No new pattern headache complaint
* No recent whiplash injury (within 3 mo)
* No spinal fractures/dislocations
* No disc problems with radiating symptoms to the arms or legs
* No severe degenerative joint disease in the spine
* No connective tissue disorders
* No primary fibromyalgia
* No metabolic or metaplastic bone disease
* No diagnosed condition that causes fainting during postural changes, such as POTS or orthostatic hypotension
* No history of cervical, thoracic, or lumbar spine surgery
* No uncontrolled high blood pressure or vascular disease
* No current use of anticoagulant therapy
* No current use of short-acting benzodiazepines, including midazolam & triazolam
* No change in medications in the past 6 weeks or intentions to change medications during the study
* Inability to walk unassisted on a treadmill
* No pacemakers or known heart conditions that influence the electrical or mechanical function of the heart, such as severe heart valve disease
* Not a DC or a DC student enrolled 4th quarter or above
* No present, self-reported pregnancy
* No chiropractic care in the 2 weeks prior to participation
* Did not participate in the feasibility study for this pilot (Perceptions and experiences following a single session of simulated or genuine high velocity, low amplitude (HVLA) manual chiropractic adjustments)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Participant blinding | Immediately post-session 1 (day 1)
  The blinding index is scaled to an internal of -1 to +1, +1 being complete lack of blinding, 0 being consistent with perfect blinding, -1 indicating opposite guessing which may be related to unblinding.
Participant blinding | Immediately pre-session 2 (day 2)
  The blinding index is scaled to an internal of -1 to +1, +1 being complete lack of blinding, 0 being consistent with perfect blinding, -1 indicating opposite guessing which may be related to unblinding.
Participant blinding | Immediately post-session 2 (day 2)
  The blinding index is scaled to an internal of -1 to +1, +1 being complete lack of blinding, 0 being consistent with perfect blinding, -1 indicating opposite guessing which may be related to unblinding.

SECONDARY OUTCOMES:
High-frequency Heart Rate Variability (HF-HRV) | baseline
  3 sensors on torso. HF-HRV indexes fluctuations in the heart period that occur within the 0.12 to 0.5 Hz frequency range
High-frequency Heart Rate Variability (HF-HRV) | post-session 2 (day 2)
  3 sensors on torso. HF-HRV indexes fluctuations in the heart period that occur within the 0.12 to 0.5 Hz frequency range.
Pre-ejection period (PEP) | baseline
  3 ECG sensors on the torso + 4 ICG sensors (2 sensors on chest and 2 sensors on back). The PEP is the time interval between the electrical depolarization of the heart (Q-wave on ECG) and the beginning of blood ejection from the heart (B-point on ICG).
Pre-ejection period (PEP) | post-session 2 (day 2)
  3 ECG sensors on the torso + 4 ICG sensors (2 sensors on chest and 2 sensors on back). The PEP is the time interval between the electrical depolarization of the heart (Q-wave on ECG) and the beginning of blood ejection from the heart (B-point on ICG).
The speed of the participants will be assessed at baseline as part of the gait analysis. | baseline
  16 inertial measurement unit (IMU) sensors (noraxon) and treadmill output measurements
The speed of the participants will be assessed again at post-session 2 as part of the gait analysis. | post-session 2 (day 2)
  16 inertial measurement unit (IMU) sensors (noraxon) and treadmill output measurements
Force measurements generated during walking will be assessed at baseline as part of the gait analysis. | baseline
  16 inertial measurement unit (IMU) sensors (noraxon) and treadmill output measurements
Force measurements generated during walking will be assessed again at post-session 2 as part of the gait analysis. | post-session 2 (day 2)
  16 inertial measurement unit (IMU) sensors (noraxon) and treadmill output measurements
Gait symmetry will be assessed at baseline as part of the gait analysis. | baseline
  16 inertial measurement unit (IMU) sensors (noraxon)
Gait symmetry will be assessed again at post-session 2 as part of the gait analysis. | post-session 2 (day 2)
  16 inertial measurement unit (IMU) sensors (noraxon)
Root Mean Square of Successive Differences (RMSSD) | baseline
  3 sensors on torso. RMSSD is a measure of heart rate variability (HRV) that focuses on short-term beat-to-beat changes in the heart period.
Root Mean Square of Successive Differences (RMSSD) | post-session 2 (day 2)
  3 sensors on torso. RMSSD is a measure of heart rate variability (HRV) that focuses on short-term beat-to-beat changes in the heart period.

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, DC, PhD, Principal Investigator — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No